CLINICAL TRIAL: NCT00658710
Title: Impact of Prolonged Physical Therapy on Gait Performance of Chronic Phase Stroke Patients
Acronym: HEMIMARCHE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0701040; 2007-A00747-46
Record Dates: First submitted 2008-04-11; First posted 2008-04-15 (Estimated); Last update posted 2013-11-07 (Estimated); Status verified 2013-11

CONDITIONS: Hemiplegia
Keywords: hemiplegia; stroke; TRIDENT
MeSH Terms: conditions — Hemiplegia; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): patients who continue physical therapy sessions during two months.
  Interventions: Behavioral: physical therapy sessions
- 2 (No Intervention): patients who stop physical therapy sessions during two months

INTERVENTIONS:
Behavioral: physical therapy sessions — two physical therapy sessions per week for two months
  Arms: 1

SUMMARY:
The aim of this multi-center, randomized controlled study is to acquire and compare information on gait performance in patients with chronic hemiplegia (six months to two years post-stroke) who either continue to attend two physical therapy sessions per week for two months or who stop physical therapy sessions for two months.Following the initial screening, subjects will be randomized into two groups: one who continues attending two physical therapy sessions per week for two months, or the other one who stops physical therapy sessions for two months. Before and after those two months, a 3 days recording will be made using an ambulatory system called TRIDENT.

DETAILED DESCRIPTION:
The aim of this multi-center, randomized controlled study is to acquire and compare information on gait performance in patients with chronic hemiplegia (six months to two years post-stroke) who either continue to attend two physical therapy sessions per week for two months or who stop physical therapy sessions for two months. This will permit us 1) to assess the efficacy of continuing physical therapy sessions during the chronic phase of post-stroke hemiplegia, 2) to investigate whether the effects of physical therapy in these patients gradually decreases during the period of six months to two years post-stroke, and 3) to model the relationship between standard measures of gait performance (speed, endurance, balance, use of technical aids…) with other multidimensional covariates: social and environmental factors (type of housing, presence of a third person,…), cognitive factors (cognitive disorders associated) and thymic factors (anxiety, depression) and 4) to assess the costs associated with the physical therapy care of chronic-phase stroke patients .

ELIGIBILITY:
Inclusion Criteria:

* Patients must be aged 18 to 75 years, with a first ischemic or hemorrhagic stroke at least six months ago and no longer than two years ago, without subsequent stroke. It must have caused initially complete hemiplegia of the right or left hemibody, but they must be able of walk alone with or without technical assistance over a distance of at least 10 meters They must be able change direction too.
* Finally, they must have a Functional Ambulation Classification (FAC) score between 4 and 6 during the inclusion.

Exclusion Criteria:

* We will exclude patients with a neurological history other than a stroke, a psychiatric illness, or an associated debilitating disease.
* They must not have an associated cerebella syndrome or a clinical brainstem attack.
* We will refuse patients who are pregnant, who have not signed the written consent, and who aren't entitled to a social security scheme.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2008-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
the average number of steps per day recorded over 3 days in an outpatient setting | day 3 and then 6 months later

SECONDARY OUTCOMES:
the scores to the scales (the 6 minutes walking test, the Wade's test, the Rivermead Mobility Index Score, the Barthel Index Score) | day 0 and then day 55
for the medico-economic study, the direct medical and non-medical costs associated with physical therapy of chronic stroke patients | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Giraux, MD, Principal Investigator — CHU ST Etienne
Locations (5):
- France (5):
  - Centre Régional de Réeducation et de Réadaptation Fonctionnelle, Angers
  - Groupe hospitalier Pellegrin CHU Bordeaux, Bordeaux
  - Hôpital J. Rebeyrol, Limoges
  - Institut Régional de médecine physique et de Réadaptation, Nancy
  - CHU de St Etienne, Saint-Etienne